CLINICAL TRIAL: NCT04740086
Title: "Feasibility and Safety of the Calcium Alginate Hydrogel Sealant for the Treatment of Cryptoglandular Fistula-in-ano"
Brief Title: "Feasibility and Safety of the Calcium Alginate Hydrogel Sealant for the Treatment of Cryptoglandular Fistula-in-ano: Phase I/IIa Clinical Trial"
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: HAS15
Record Dates: First submitted 2021-01-21; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-01

CONDITIONS: Anal Fistula
Keywords: cryptoglandular anal fistula; calcium alginate; sealant
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Calcium alginate hydrogel — 1. The external and internal fistulous orifice and fistulous tract were explored without applying any product, including hydrogen peroxide or povidone-iodine.
  2. The seton was removed and FT cannulation was performed using a needle for cleaning with a gauze impregnated with saline.
  3. Calcium chloride was applied through the EFO until it exits through the IFO, and then the IFO was obturated.
  4. Alginate was applied, and the pressure at the IFO was stopped, until the alginate solution partial exits through the IFO.
  5. The IFO was closed with a 3/0 braided resorbable suture.
  6. The EFO was removed with an electric scalpel and closed with a 3/0 braided resorbable suture.

SUMMARY:
Background: Complex perianal fistulas pose a challenge to surgeons since the fistulous tract must be eliminated without impairing continence. Biological sealants have emerged as an effective alternative for maintaining the integrity of the anal sphincter. The investigators aimed to assess the feasibility and safety of calcium alginate hydrogel injections into the tract as treatment for complex cryptoglandular fistulas.

Methods: A prospective, single-center, case series of this novel technique was conducted in a level 3 hospital, including patients diagnosed with trans-sphincteric perianal fistulas and treated with a calcium alginate hydrogel sealant. A strict follow-up was performed by an independent surgeon at 1, 3, 6, and 12 months. The main outcome measures were feasibility, safety (number of adverse events) and efficacy of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age ≥18 years
* Cryptoglandular PAF treated by Seton placement for at least 3 months, with a single External Fistulous Orifice and Internal Fistulous Orifice

Exclusion Criteria:

* Informed Consent Form not signed or withdrawn
* Not possible to adhere to follow-up routine
* Another investigational drug in the previous 3 months
* Allergy to alginate
* Grade IV in American Society of Anesthesiologists scale
* Pregnancy
* History of radiotherapy in the perineal area
* Diagnosis or suspicion of Intestinal Blow Disease
* Immunosuppression, active neoplasia at the time of recruitment or in previous year, or positive for human immunodeficiency virus Internal Fistulous Orifice not located during the procedure
* Simple anal fistula (submucosa or low Intersphincteric Perianal Fistula, except association with Faecal Incontinence
* Anal stenosis that prevents exploration
* Undrained collections >2 cm
* Rectovaginal fistulas
* Fistulas of non-cryptoglandular origin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients with a single complex cryptoglandular perianal fistula
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-01-01; Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of patients treated following the protocol during the surgery | During the surgery
  Feasibility is measured as the ratio between the number of patients who received the injection following all the steps of the protocol and the total number of individuals included in the study.
Incidence of adverse events at 1 month | At 1 month
  Incidence of adverse events, their relationship to the product under investigation, and their intensity (mild, moderate, or severe)
Incidence of adverse events at 3 months | At 3 months
  Incidence of adverse events, their relationship to the product under investigation, and their intensity (mild, moderate, or severe)
Incidence of adverse events at 6 months | At 6 months
  Incidence of adverse events, their relationship to the product under investigation, and their intensity (mild, moderate, or severe)
Incidence of adverse events at 12 months | At 12 months
  Incidence of adverse events, their relationship to the product under investigation, and their intensity (mild, moderate, or severe)

SECONDARY OUTCOMES:
Ecographic curation at 12 months | At 12 months
  Closure of the external fistulous orifice that prevented the injection of hydrogen peroxide diluted to 50 percent, in addition to the absence of hyperechogenic collections and images suggesting the existence of pus or air in the tract.
Clinical curation at 1 month | At 1 month
  Complete cure defined as the absence of suppuration and scarring in the external fistulous orifice; partial cure defined as the absence of suppuration and scarring in the external fistulous orifice without complete re-epithelialization; treatment failure or lack of cure defined as suppuration and/or scarring in the external fistulous orifice
Clinical curation at 3 months | At 3 months
  Complete cure defined as the absence of suppuration and scarring in the external fistulous orifice; partial cure defined as the absence of suppuration and scarring in the external fistulous orifice without complete re-epithelialization; treatment failure or lack of cure defined as suppuration and/or scarring in the external fistulous orifice
Clinical curation at 6 months | At 6 months
  Complete cure defined as the absence of suppuration and scarring in the external fistulous orifice; partial cure defined as the absence of suppuration and scarring in the external fistulous orifice without complete re-epithelialization; treatment failure or lack of cure defined as suppuration and/or scarring in the external fistulous orifice
Clinical curation at 12 months | At 12 months
  Complete cure defined as the absence of suppuration and scarring in the external fistulous orifice; partial cure defined as the absence of suppuration and scarring in the external fistulous orifice without complete re-epithelialization; treatment failure or lack of cure defined as suppuration and/or scarring in the external fistulous orifice

CONTACTS AND LOCATIONS:
Locations (1):
- Sandra Dios Barbeito, Seville, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de la Portilla F, Dios-Barbeito S, Maestre-Sanchez MV, Vazquez-Monchul JM, Garcia-Cabrera AM, Ramallo I, Reyes-Diaz ML. Feasibility and safety of calcium alginate hydrogel sealant for the treatment of cryptoglandular fistula-in-ano: phase I/IIa clinical trial. Colorectal Dis. 2021 Jun;23(6):1499-1506. doi: 10.1111/codi.15608. Epub 2021 Mar 20. PMID 33655675